CLINICAL TRIAL: NCT00006021
Title: Phase I/II Trial of Arsenic Trioxide (As2O3) With Ascorbic Acid in the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Arsenic Trioxide Plus Vitamin C in Treating Patients With Recurrent or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20000156; CDR0000068033 (Registry Identifier: PDQ (Physician Data Query)); SCCC-2000010 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Ascorbic Acid; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: ascorbic acid
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Vitamin C may increase the effectiveness of arsenic trioxide by making cancer cells more sensitive to the drug.

PURPOSE: Phase I/II trial to determine the effectiveness of arsenic trioxide plus vitamin C in treating patients who have recurrent or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of arsenic trioxide when administered with ascorbic acid in patients with recurrent or refractory multiple myeloma.
* Determine the therapeutic efficacy of this treatment combination in these patients.
* Determine the expression of MDR and Bcl-xL genes and the intracellular levels of GSH in these patients before and after this treatment regimen and assess whether these measures have prognostic value.

OUTLINE: This is a multicenter, dose-escalation study of arsenic trioxide.

* Phase I: Patients receive arsenic trioxide IV over 1-4 hours and ascorbic acid IV over 5-10 minutes on days 1-5 weekly for 5 weeks. Treatment continues every 7 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive the MTD of arsenic trioxide with ascorbic acid as outlined above.

Patients are followed monthly for up to 5 years.

PROJECTED ACCRUAL: A total of 31-43 patients (6-18 for phase I and 16-25 for phase II) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma

  * M-protein by serum protein electrophoresis or urine protein electrophoresis
  * Quantitative determination of immunoglobulin
  * Bone marrow biopsy and aspirate with a plasma cell count greater than 10%
  * Refractory or chemoresistant disease defined as failure to respond (less than 50% reduction in M protein level) or progression within 2 months after receiving at least 2 chemotherapy regimens including:

    * Alkylating based regimen (melphalan) in combination with steroids (prednisone) or other chemotherapy regimens (e.g., vincristine, bleomycin, melphalan, cyclophosphamide, and prednisone or vincristine, carmustine, doxorubicin, and prednisone)
    * Vincristine, doxorubicin, and dexamethasone (VAD) regimen
    * Pulse therapy with high dose steroids alone
    * High dose alkylating agent and autologous stem cell transplantation
    * Allogeneic bone marrow transplantation
  * Plateau phase defined as M protein in the serum or urine for more than 6 weeks despite response to prior therapy

    * Must have received at least 2 of the chemotherapy regimens listed above or equivalent regimens
  * Recurrent disease defined as progression more than 2 months after initial therapy and failure to respond (less than 50% reduction or progression in M protein levels) to 1 chemotherapy regimen listed above or other salvage regimens (e.g., high-dose cyclophosphamide or topotecan)

    * Must have received VAD or other equivalent chemotherapy regimen
    * Should be considered for autologous or allogenic transplantation
    * Prior local radiotherapy allowed

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3*
* Platelet count at least 50,000/mm^3* NOTE: *Unless attributable to bone marrow infiltration by multiple myeloma

Hepatic:

* Bilirubin less than 3 mg/dL
* Transaminases less than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine less than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No cardiac arrhythmias including recurrent supraventricular arrhythmia, any type of sustained ventricular arrhythmia, or conduction block (atrioventricular block grade II or III, left bundle branch block)
* Ejection fraction at least 30%
* No uncontrolled ischemic heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 4 months after study
* HIV negative
* No grade 3 or higher neurological disorder, including seizure disorders
* No underlying medical condition that would preclude study
* No other active malignancy except adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 2 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* Concurrent steroid treatment allowed except for primary treatment of myeloma

Radiotherapy:

* See Disease Characteristics
* Concurrent local radiotherapy for pain or symptom control allowed provided the pain or symptom is not related to disease progression

Surgery:

* Not specified

Other:

* No other concurrent ascorbic acid supplements
* No other concurrent investigational drug or therapy
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-06; Primary Completion 2006-05 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Disease response as measured by M protein quantitation and the percentage of plasma cell infiltration in bone marrow biopsies after every course

SECONDARY OUTCOMES:
Toxicity as measured by CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lee, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Cedars Medical Center, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center at Mount Sinai Medical Center, Miami Beach, Florida

REFERENCES:
- [Result] Bahlis NJ, McCafferty-Grad J, Jordan-McMurry I, Neil J, Reis I, Kharfan-Dabaja M, Eckman J, Goodman M, Fernandez HF, Boise LH, Lee KP. Feasibility and correlates of arsenic trioxide combined with ascorbic acid-mediated depletion of intracellular glutathione for the treatment of relapsed/refractory multiple myeloma. Clin Cancer Res. 2002 Dec;8(12):3658-68. PMID 12473574